CLINICAL TRIAL: NCT02284867
Title: Comparison Between Uterine Natural Killer Cells In Preterm Labor And Term Labor
Brief Title: Are Uterine Natural Killer Cells Involved in the Initiation of Preterm Labor ?
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Abass, Assistant lecturer, Ain Shams University
Other Study IDs: NK Cells & Pretem labor; preterm labor pathogenesis (Other: AinShamsU)
Record Dates: First submitted 2014-11-02; First posted 2014-11-06 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Preterm Labour
Keywords: uterine natural killer cells; CD16; CD56; Preterm labour
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — a placental sample will be taken either the patient delivered preterm or at term (term patients will be either control term group or patients with successful treatment of preterm labor). The placental sample taken should have part of the decidua and then the sample will be fixed in 10% neutral-buffered formalin for 24-48 h, routinely processed, embedded in paraffin wax, sectioned at 3 μm thickness, and mounted on 3-aminopropyl-triethoxysilane -coated slides. Serial sections will be immunostained for CD 16 and CD56 . Immunohisto-chemistery study will be done at Ain Shams Maternity Hospital Histopathology department.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preterm labor: Patients who has threatened preterm labor and will receive tocolysis and these patients will either not respond to tocolysis and delivered preterm or will respond to tocolysis and will deliver at term .
  Interventions: Other: immunohistochemistry study
- Term labor: Patient delivered vaginally at term with no history of having tocolysis for preterm labor at the current pregnancy .
  Interventions: Other: immunohistochemistry study

INTERVENTIONS:
Other: immunohistochemistry study — After taking informed written consent,a placental sample will be taken either the patient delivered preterm or at term (term patients will be either control term group or patients with successful treatment of preterm labor). The placental sample taken should have part of the decidua and then the sample will be fixed in 10% neutral-buffered formalin for 24-48 h, routinely processed, embedded in paraffin wax, sectioned at 3 μm thickness, and mounted on 3-aminopropyl-triethoxysilane -coated slides. Serial sections will be immunostained for CD 16 and CD56 . immunohistochemistry study will be done at Ain Shams Maternity Hospital Histopathology department.

SUMMARY:
Research question:

Population of study: women diagnosed as term pregnancy in labor (control) and the other group diagnosed as preterm labor (cases).

Intervention: measuring uterine natural killer cells . Outcome: uterine natural killer cells has a role in initiation of preterm labor.

Research hypothesis:

• Are uterine Natural Killer cells involved in the initiation of preterm labor ?

Medical Application:

• Possibility of prediction of preterm labor by assessment of Natural killer cells as well as preventing preterm labor by suppressing their activity .

DETAILED DESCRIPTION:
Type of the Study:

This is a case control study .

Study Settings:

This clinical trial will be conducted at Ain Shams University Maternity Hospital and the laboratory work will be done at Ain Shams University histopathology Laboratory , in the period between August 2012 to August 2014 .

Study Population:

The patients will be recruited from women attending casualty at Ain Shams University Maternity Hospital.

The included patients will be

Divided into two groups:

* Group 1: Patients who has threatened preterm labor and will receive tocolysis and these patients will either not respond to tocolysis and delivered preterm or will respond to tocolysis and will deliver at term .
* Group 2: Patient delivered vaginally at term with no history of having tocolysis for preterm labor at the current pregnancy .

Intervention:

After taking informed written consent, the recruited patients will be subjected to the following:

- History taking, with particular emphasis on: Past medical history (no diabetes mellitus, no hypertension, etc..) Past obstetric history (history of preterm labor). Menstrual history(to be sure of her LMP( last menstrual period) and this date is reliable).

* Having earlier ultrasound to document gestational age.
* History of labor pains which is becoming regular and frequent.
* No suggestive history of preterm prelabor rupture of membranes
* General examination with particular emphasis on blood pressure, weight and height.
* Abdominal examination with particular emphasis on uterine activity.
* Obstetric ultrasound (transabdominal) to document viability of pregnancy and to ensure the gestational age.
* Included patients will receive tocolysis (according to Ain Shams University Maternity hospital protocol which is recommending usage of calcium channel blocker (Nifedipine) Initially 10mg orally every 15 minutes, up to 4 doses of Nifedipine to stop contractions. After this slow release nifedipine. It has been found that an 8 hourly dosage of 40mg - 20mg - 40mg calcium channel blocker is suitable for most women. This is in addition to use of steroids to enhance lung maturity (dexamethasone, 6 mg intramuscular /12 hrs for 48 hrs)
* Patients will be traced by fetal monitor and uterine tocodynamometer (Oxford Sonicaid Team ®)to monitor uterine contractions and if the treatment was successful or not.
* After delivery a placental sample will be taken either the patient delivered preterm or at term (term patients will be either control term group or patients with successful treatment of preterm labor). The placental sample taken should have part of the decidua and then the sample will be fixed in 10% neutral-buffered formalin for 24-48 h, routinely processed, embedded in paraffin wax, sectioned at 3 μm thickness, and mounted on 3-aminopropyl-triethoxysilane -coated slides. Serial sections will be immunostained for CD 16 and CD56 . immunohistochemistry study will be done at Ain Shams Maternity Hospital Histopathology department.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age: 18-35 years old (to decrease the incidence of preterm labor related to age factor).
2. Women who present with viable pregnancy (between 28 and 37 weeks' gestation), and having a threatened preterm labor (which is defined as ≥ 2 uterine contractions at 28-37 weeks' gestation, The onset of labor may be determined by documented uterine contractions (at least one every 10 minutes) and ruptured fetal membranes or documented cervical change with an estimated length of less than 1cm or cervical dilation of more than 2 cm. Threatened preterm labor may be diagnosed when there are documented uterine contractions but no evidence of cervical change.

Exclusion Criteria:

1. Multiple pregnancy.
2. Documented uterine anomalies.
3. Oligohydramnios and polyhydramnios .
4. Medical disorders as Diabetes mellitus and hypertension.
5. Preterm premature rupture of membranes.
6. Conditions that may have an influence on immune reaction e.g. history of chorioamnionitis.
7. Smoking as a risk factor for preterm labor.
8. Patients having Autoimmune disorder as it may affect Uterine NK( natural killer ) cells level .

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The patients will be recruited from women attending casualty at Ain Shams University Maternity Hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murad Elsaed, proffesor, Study Chair — +02-01223165820

REFERENCES:
- [Background] Koga K, Cardenas I, Aldo P, Abrahams VM, Peng B, Fill S, Romero R, Mor G. Activation of TLR3 in the trophoblast is associated with preterm delivery. Am J Reprod Immunol. 2009 Mar;61(3):196-212. doi: 10.1111/j.1600-0897.2008.00682.x. PMID 19239422
- [Background] Murphy SP, Hanna NN, Fast LD, Shaw SK, Berg G, Padbury JF, Romero R, Sharma S. Evidence for participation of uterine natural killer cells in the mechanisms responsible for spontaneous preterm labor and delivery. Am J Obstet Gynecol. 2009 Mar;200(3):308.e1-9. doi: 10.1016/j.ajog.2008.10.043. Epub 2008 Dec 27. PMID 19114277

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Our study was conducted at Ain Shams University Maternity Hospital during the period between August 2012 and December 2014. A total of 60 pregnant women were included in the study.
Pre-assignment Details: Adequate placental tissue sampled and proper primary storage technique then proper way of staining
Period: Overall Study
Arm/Group | Preterm Labor | Term Labor
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preterm Labor | Term Labor | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (4) | 26.4 (3.9) | 26.1 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Parity [Median (Inter-Quartile Range); unit: live birth] | 1 [0 to 1] | 2 [1 to 2] | 1 [0 to 2]
Body Mass Index [Mean (Standard Deviation); unit: Kg/M^2] | 21.7 (2.3) | 21.8 (2.3) | 21.7 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Uterine Natural Killer Cells In Preterm Labor
Description: Number of participants with CD16 orCD 56 uterine Natural Killer Cells positive staining of placental sample
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Preterm Labor | Term Labor
Number analyzed (Participants) | 30 | 30
participants
  CD16+ uterine Natural Killer Cells | 21 | 1
  CD56 bright uterine Natural Killer cells | 0 | 0
Statistical Analysis 1: Comparison: Preterm Labor vs Term Labor; Categorical data were presented as number and percentage and differences were compared using the Pearson chi-squared test. Ordinal data were compared using the chi-squared test for trend A two-sided p-value <0.05 was considered statistically significant; Test type: Non-Inferiority or Equivalence — Multivariable binary logistic regression was done to examine the relation between CD16+ NK and preterm labor as adjusted for other confounding factors the enter method was used to build the regression model. A two-sided p-value <0.05 was considered statistically significant; p < 0.0002, Regression, Logistic — To our best of known , no previous human studies was analyzing this issue; Odds Ratio (OR) = 65.01, 95% CI 2-sided [6.96 to 606.76], Standard Error of Mean 1.14

2. Secondary Outcome: Comparison of CD16+ CD56 Dim Uterine Natural Killer Cells (uNK) Prevalence in Decidua vs. Villi in Placenta of Both Study Groups
Description: CD16+ CD56dim uterine Natural Killer cells (uNK) in the villi was found in Preterm delivery Group.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Preterm Labor | Term Labor
Number analyzed (Participants) | 30 | 30
participants
  Positive CD16+ CD56 dim villous only NK cells | 1 | 10
  Positive CD16+ CD56dim villos and decidua NK cells | 0 | 11

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Preterm Labor | Term Labor
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No